CLINICAL TRIAL: NCT04392544
Title: Interrogation of the Prevalence of Intestinal Inflammation in Cystic Fibrosis Patients and the Correlation with Abdominal Symptoms
Brief Title: Intestinal Inflammation in CF Patients
Status: Active, not recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Tanja Gonska, Associate Professor and Senior Associate Scientist, The Hospital for Sick Children
Other Study IDs: 1000060079
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis in Children; Cystic Fibrosis Gastrointestinal Disease; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples to assess Calprotectin levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pediatric: Pediatric CF population age 10-18 years.
- Adult: Adult CF population age ≥ 18 years.

SUMMARY:
Cystic Fibrosis (CF) is a disease that affects salt and water transport in multiple organs. Many CF patients suffer from abdominal pain and this could be due to intestinal inflammation. However, so far we do not know how many of the CF patients actually do have intestinal inflammation when looking at intestinal specimens. There is a proven connection between chronic inflammation and developing colorectal cancer and over the years more CF patients are developing colorectal cancer. Thus, it becomes increasingly important to look for the presence of intestinal inflammation in CF patients since early treatment may improve their symptoms and reduce the risk for colorectal cancer.

DETAILED DESCRIPTION:
The aim is to determine the prevalence of intestinal inflammation by measurement of fecal calprotectin and/or histological evaluation of intestinal tissue biopsies in both pediatric and adult CF populations.

Pediatric CF population (Age 10-18 years):

1. Determine the prevalence of intestinal inflammation in a cohort of pediatric CF patients based on fecal calprotectin levels in stool samples.
2. Assess the correlation between fecal calprotectin and abdominal symptoms/QOL.

Adult CF population (Age ≥ 18 years):

1. Determine the prevalence of intestinal inflammation in a cohort of adult CF patients based on histological evaluation of intestinal tissues biopsies and fecal calprotectin levels in stool samples

   1. in adult CF patients who have not undergone lung or liver transplantation.
   2. in adult CF patients who have undergone lung or liver transplantation.
2. Assess the correlation between fecal calprotectin and histological-proven intestinal inflammation in adult CF patients.
3. Assess the correlation between histological-proven intestinal inflammation and abdominal symptoms/QOL as well as the correlation between fecal calprotectin and abdominal symptoms/QOL.

ELIGIBILITY:
INCLUSION CRITERIA ;

Pediatric cohort:

1. Diagnosis of CF
2. Informed consent obtained
3. Age 10-18 years

Adult cohort:

1. Diagnosis of CF
2. Informed consent obtained
3. Age ≥ 18 years
4. Patient undergoing a colonoscopy for a clinical indication

EXCLUSION CRITERIA ;

Pediatric Cohort:

1. Patients with the diagnosis of IBD.
2. Patients during an episode of acute gastroenteritis or a pulmonary exacerbation.

Adult cohort:

1. Patients with the diagnosis of IBD.
2. Any health condition, e.g. coagulopathy, sepsis, severe bacterial colitis that would increase the risk for perforation or bleeding when taking intestinal tissue biopsies.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult population diagnosed of cystic fibrosis will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure fecal calprotectin levels in stool samples of CF pediatric population to determine prevalence of intestinal inflammation. | Day 1
Assess the correlation between fecal calprotectin levels and abdominal symptoms. | Day 1
Determine the prevalence of intestinal inflammation in adult CF patients based on histological evaluation of intestinal tissues biopsies and fecal calprotectin levels in stool samples. | Day 1
  Sub groups; with and without lung or liver transplantation.
Determine the correlation between fecal calprotectin and histological-proven intestinal inflammation in adult CF patients. | Day 1
Assess the correlation between histological-proven intestinal inflammation and abdominal symptoms in adult CF patients. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Gonska, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada